CLINICAL TRIAL: NCT02111746
Title: A Prospective Randomized-controlled Study on Effectiveness of Extended-release Liposomal Bupivacaine in Postoperative Pain Control
Brief Title: PAIN - Postoperative Analgesia INvestigation
Acronym: PAIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Kristofer Charlton-Ouw, Associate Professor, Department of Cardiothoracic and Vascular Surgery, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTVS-KC02; HSC-MS-13-0620 (Other: UTHSC IRB); NCT02474472 (obsolete NCT alias)
Record Dates: First submitted 2014-04-02; First posted 2014-04-11 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; sternotomy; laparotomy; thoracotomy; mini-thoracotomy; truncal surgical incisions; local anaesthetics; bupivacaine
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Analgesia, Patient-Controlled

STUDY DESIGN:
Intervention Model Description: Prospective, blinded, controlled randomized clinical trial with 2-armed parallel-group sequential design
Who Masked: Participant, Investigator
Masking Description: Masking included all patients, who were blinded to the contents of the intraoperative injection, as well as partial blinding of the surgical team who were masked from the treatment allocation up until the time of injection following which the knowledge of drug was inevitable as Exparel® has a milky appearance as opposed to the colorless bupivacaine hydrochloride (standard) formulations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exparel® (Experimental): Patients in this group will receive will receive the study drug [bupivacaine liposomal injectable suspension (Exparel®)] and Patient Controlled Analgesia (PCA). Exparel® is an FDA-approved bupivacaine liposome injectable suspension produced by Pacira Pharmaceuticals.
  Interventions: Drug: Exparel; Drug: Patient Controlled Analgesia (PCA)
- Regular Bupivacaine (Active Comparator): Patients in this group will receive will receive the standard regular bupivacaine hydrochloride (HCl) and PCA. Bupivacaine HCl is an FDA-approved injectable suspension. The standard non-liposomal bupivacaine will be from Hospira pharmaceuticals
  Interventions: Drug: Bupivacaine hydrochloride; Drug: Patient Controlled Analgesia (PCA)

INTERVENTIONS:
Drug: Exparel — Participants will receive 266mg of liposomal bupivicaine (equivalent of one 1.3% 20ml vial of EXPAREL®) diluted in 60ml of preservative-free normal (0.9%) sterile saline for a total volume of 80mL. Drug will be administered at the end of the procedure just prior to wound closure.
  Other Names: bupivacaine liposomal injectable suspension (Exparel®)
  Arms: Exparel®
Drug: Bupivacaine hydrochloride — Participants will receive 125mg of bupivacaine hydrochloride (equivalent of one 0.25% 50ml or five 0.25% 10ml vials ) diluted in 30ml of preservative-free normal (0.9%) sterile saline for a total volume of 80mL. Drug will be administered at the end of the procedure just prior to wound closure.
  Other Names: Regular Bupivacaine
  Arms: Regular Bupivacaine
Drug: Patient Controlled Analgesia (PCA) — Patients will have access to the standard Patient Controlled Analgesia (PCA) offered at the Memorial Hermann Hospital - Texas Medical Center. The PCA drug will be Dilaudid (hydromorphone). Initial dosing will be per the standard hospital protocol of 0.2 mg demand dose, 10 minute lockout, 2 mg per hour max, 0.4 mg rescue dose. Adjustments to the PCA dosing will be made based on clinical needs. Patients will receive PCA until the third postoperative day

SUMMARY:
The purpose of this study is to assess the efficacy of the intraoperative injection of prolonged acting (liposomal) bupivacaine in postoperative pain control after truncal surgical incisions.

DETAILED DESCRIPTION:
Study Design:

This is a prospective, single-institution, parallel-group, single-blinded, randomized-controlled, two-arm, effectiveness study comparing bupivacaine liposomal injectable suspension (Exparel®) versus regular bupivacaine hydrochloride (HCl).

Procedure:

In patients aged 18 and over who require sternotomy, thoracotomy, mini-thoracotomy, or laparotomy incisions will be screened and consented for potential enrollment. Patients will be randomized following consenting to either Exparel® or regular bupivacaine hydrochloride group.

Course of Study:

The study will accrue patients over the course of 4 years.

Enrollment:

Enrollment will consist of all adult patients aged 18 and over undergoing surgical procedures requiring sternotomy, thoracotomy, mini-thoracotomy, or laparotomy incisions. Patients will be screened and consented preoperatively. If the patient is deemed eligible and consents to participate, randomization will occur and the patient will be considered enrolled.

Recruitment:

The target for enrollment will be 280 patients (the study target sample size per power analysis, but actual enrollment will be greater (330 patients) to account for exclusions for various reasons in order to achieve the target recruitment).

Risks:

There is a small increased risk to the patients by participating in the study in addition to a possible chance of breach in patient confidentiality as the study involves evaluation of an FDA-approved drug. As detailed in the informed consent, the subjects are at risk of developing adverse effects from Exparel®, described on the drug packet insert and from HCl Bupivacaine, also described on the drug packet insert. The investigators do not expect any additional physical risks other than an unintentional disclosure of sensitive patient health information.

Data Safety Monitoring:

As the Principal Investigator of this study, Dr. Charlton-Ouw from the Department of Cardiothoracic and Vascular Surgery at The University of Texas at Houston Medical School will conduct the data safety monitoring of this study. He will annually meet with all other co-investigators to review the patients enrolled in this study. As part of the data safety monitoring plan, all patients enrolled until that point in time would be unblinded in order to review the outcomes. Additionally, in view of the uncertainty attached to the treatment effects in this heterogeneous population, owing to limited currently available data, an independent Data Safety Monitoring Committee, will oversee the progress of the trial.

IND#:

The drugs that will be used are already approved by the FDA and do not have IND/IDE#

Proposed Funding Source:

The study is internally funded and is investigator-initiated.

Communication of Study Results:

The communication of study results will occur only between authorized individuals who are listed to take part in the study through our department. The individuals who will take part in the study will acknowledge and adhere to the importance of patient safety and the protection of their private information. The results of this study will be analyzed and published after the approval of the principal investigator, co-investigators, and biostatistician in a peer-reviewed scientific journal and/or presented at an international/national scientific conference or meeting regardless of outcome.

ELIGIBILITY:
Inclusion Criteria:

* 18 years-old or older, and
* Sternotomy, thoracotomy, laparotomy or mini-thoracotomy incision is planned
* There is reasonable expectation that the patient will be extubated within 24 hours after surgery

Exclusion Criteria:

* The patient has a known allergy to morphine or any opioid
* The patient has a known chronic pain disorder or takes daily opioid medication > 1 month prior to surgery
* There is anticipated difficulty communicating pain status due to language or other barriers at the investigator discretion
* High postoperative morbidity index based on preoperative assessment, such as, low likelihood of extubation within 24 hours, extensive thoracoabdominal aortic aneurysm (Extent 2 TAAA), preoperative renal insufficiency/failure, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2013-11-20 (Actual); Primary Completion 2017-05-03 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristofer M Charlton-Ouw, MD FACS, Principal Investigator — University of Texas Health Science Center, Department of Cardiothoracic and Vascular Surgery, UT Medical School at Houston
Locations (1):
- Department of Cardiothoracic and Vascular Surgery and Memorial Hermann Heart and Vascular Institute - Texas Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sandhu HK, Miller CC 3rd, Tanaka A, Estrera AL, Charlton-Ouw KM. Effectiveness of Standard Local Anesthetic Bupivacaine and Liposomal Bupivacaine for Postoperative Pain Control in Patients Undergoing Truncal Incisions: A Randomized Clinical Trial. JAMA Netw Open. 2021 Mar 1;4(3):e210753. doi: 10.1001/jamanetworkopen.2021.0753. PMID 33724391

RESULTS

PARTICIPANT FLOW:
Groups:
- Exparel®: Patients will receive will receive the study drug [bupivacaine liposomal injectable suspension (Exparel®)] and Patient Controlled Analgesia (PCA).
  Exparel: Participants will receive 266mg of liposomal bupivicaine (equivalent of one 1.3% 20ml vial of EXPAREL®) diluted in 60ml of preservative-free normal (0.9%) sterile saline for a total volume of 80mL. Drug will be administered at the end of the procedure just prior to wound closure.
  Patient Controlled Analgesia (PCA): Patients will have access to the standard Patient Controlled Analgesia (PCA) offered at the Memorial Hermann Hospital - Texas Medical Center. The PCA drug will be Dilaudid (hydromorphone). Initial dosing will be per the standard hospital protocol of 0.2 mg demand dose, 10 minute lockout, 2 mg per hour max, 0.4 mg rescue dose. Adjustments to the PCA dosing will be made based on clinical needs. Patients will receive PCA until the third postoperative day
- Regular Bupivacaine: Patients will receive will receive the standard regular bupivacaine hydrochloride (HCl) and PCA. Bupivacaine HCl is an FDA-approved injectable suspension.
  Bupivacaine hydrochloride: Participants will receive 125mg of bupivacaine hydrochloride (equivalent of one 0.25% 50ml or five 0.25% 10ml vials ) diluted in 30ml of preservative-free normal (0.9%) sterile saline for a total volume of 80mL. Drug will be administered at the end of the procedure just prior to wound closure.
  Patient Controlled Analgesia (PCA): Patients will have access to the standard Patient Controlled Analgesia (PCA) offered at the Memorial Hermann Hospital - Texas Medical Center. The PCA drug will be Dilaudid (hydromorphone). Initial dosing will be per the standard hospital protocol of 0.2 mg demand dose, 10 minute lockout, 2 mg per hour max, 0.4 mg rescue dose. Adjustments to the PCA dosing will be made based on clinical needs. Patients will receive PCA until the third postoperative day
Period: Overall Study
Arm/Group | Exparel® | Regular Bupivacaine
Started | 172 | 171
Completed | 169 | 169
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exparel® | Regular Bupivacaine | Total
Number analyzed (Participants) | 172 | 171 | 343
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age wasn't collected for all participants.
  years | 60.2 (14.8) | 61 (13.9) | 60.7 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 67 | 122
  Male | 117 | 104 | 221
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity data wasn't collected from all participants.
  Participants
    Hispanic or Latino | 27 | 26 | 53
    Not Hispanic or Latino | 139 | 132 | 271
    Unknown or Not Reported | 6 | 13 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race data wasn't collected from all participants.
  Participants
    number analyzed (Participants) | 145 | 145 | 290
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 6 | 4 | 10
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 35 | 25 | 60
    White | 98 | 103 | 201
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 6 | 13 | 19
Region of Enrollment [Number; unit: participants]
  United States | 172 | 171 | 343

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain as Assessed by a Numeric Pain Scale (NPS)
Description: The Numeric Pain Scale (NPS) ranges from 0 ("no pain") to 10 ("worst possible pain").
Time Frame: postoperative day 1
Population: Intention-to-treat analysis. Data for this measure was collected for only 153 in the Exparel arm and 152 in the Regular Bupivacaine group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exparel® | Regular Bupivacaine
Number analyzed (Participants) | 153 | 152
units on a scale | 5.05 (2.8) | 5.02 (2.68)
Statistical Analysis 1: Comparison: Exparel® vs Regular Bupivacaine; Test type: Superiority; p = 0.934, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Postoperative Pain as Assessed by a Numeric Pain Scale (NPS)
Description: The Numeric Pain Scale (NPS) ranges from 0 ("no pain") to 10 ("worst possible pain").
Time Frame: postoperative day 2
Population: Intention-to-treat analysis. Data for this measure was collected for only 160 in the Exparel arm and 159 in the Regular Bupivacaine group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exparel® | Regular Bupivacaine
Number analyzed (Participants) | 160 | 159
units on a scale | 4.69 (2.49) | 4.08 (2.64)
Statistical Analysis 1: Comparison: Exparel® vs Regular Bupivacaine; Test type: Superiority; p = 0.036, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Postoperative Pain as Assessed by a Numeric Pain Scale (NPS)
Description: The Numeric Pain Scale (NPS) ranges from 0 ("no pain") to 10 ("worst possible pain").
Time Frame: postoperative day 3
Population: Intention-to-treat analysis. Data for this measure was collected for only 159 in the Exparel arm and 151 in the Regular Bupivacaine group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exparel® | Regular Bupivacaine
Number analyzed (Participants) | 159 | 151
units on a scale | 3.71 (2.42) | 3.03 (2.47)
Statistical Analysis 1: Comparison: Exparel® vs Regular Bupivacaine; Test type: Superiority; p = 0.014, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Postoperative Pain as Assessed by a Five-point Satisfaction Scale
Description: The 5-point satisfaction scale ranges from 1 (extremely dissatisfied) to 5 (extremely satisfied).
Time Frame: postoperative day 1
Population: Intention-to-treat analysis. Data for this measure was collected for only 144 in the Exparel arm and 146 in the Regular Bupivacaine group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exparel® | Regular Bupivacaine
Number analyzed (Participants) | 144 | 146
units on a scale | 4.08 (1.16) | 3.99 (1.35)
Statistical Analysis 1: Comparison: Exparel® vs Regular Bupivacaine; Test type: Superiority; p = 0.512, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Postoperative Pain as Assessed by a Five-point Satisfaction Scale
Description: The 5-point satisfaction scale ranges from 1 (extremely dissatisfied) to 5 (extremely satisfied).
Time Frame: postoperative day 2
Population: Intention-to-treat analysis. Data for this measure was collected for only 155 in the Exparel arm and 155 in the Regular Bupivacaine group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exparel® | Regular Bupivacaine
Number analyzed (Participants) | 155 | 155
units on a scale | 4.23 (1.05) | 4.12 (1.33)
Statistical Analysis 1: Comparison: Exparel® vs Regular Bupivacaine; Test type: Superiority; p = 0.449, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Postoperative Pain as Assessed by a Five-point Satisfaction Scale
Description: The 5-point satisfaction scale ranges from 1 (extremely dissatisfied) to 5 (extremely satisfied).
Time Frame: postoperative day 3
Population: Intention-to-treat analysis. Data for this measure was collected for only 148 in the Exparel arm and 148 in the Regular Bupivacaine group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exparel® | Regular Bupivacaine
Number analyzed (Participants) | 148 | 148
units on a scale | 4.37 (0.99) | 4.37 (1.11)
Statistical Analysis 1: Comparison: Exparel® vs Regular Bupivacaine; Test type: Superiority; p = 1, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Postoperative Pain as Assessed by the Brief Pain Inventory (BPI)
Description: The Brief Pain Inventory (BPI) ranges from 0 ("no pain") to 10 ("worst pain you can imagine").
Time Frame: postoperative day 1
Population: Intention-to-treat analysis. Data for this measure was collected for only 142 in the Exparel arm and 140 in the Regular Bupivacaine group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exparel® | Regular Bupivacaine
Number analyzed (Participants) | 142 | 140
units on a scale | 5.49 (2.51) | 5.41 (2.52)
Statistical Analysis 1: Comparison: Exparel® vs Regular Bupivacaine; Test type: Superiority; p = 0.774, Wilcoxon (Mann-Whitney)

8. Primary Outcome: Postoperative Pain as Assessed by the Brief Pain Inventory (BPI)
Description: The Brief Pain Inventory (BPI) ranges from 0 ("no pain") to 10 ("worst pain you can imagine").
Time Frame: postoperative day 2
Population: Intention-to-treat analysis. Data for this measure was collected for only 151 in the Exparel arm and 149 in the Regular Bupivacaine group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exparel® | Regular Bupivacaine
Number analyzed (Participants) | 151 | 149
units on a scale | 4.48 (2.38) | 4.4 (2.5)
Statistical Analysis 1: Comparison: Exparel® vs Regular Bupivacaine; Test type: Superiority; p = 0.188, Wilcoxon (Mann-Whitney)

9. Primary Outcome: Postoperative Pain as Assessed by the Brief Pain Inventory (BPI)
Description: The Brief Pain Inventory (BPI) ranges from 0 ("no pain") to 10 ("worst pain you can imagine").
Time Frame: postoperative day 3
Population: Intention-to-treat analysis. Data for this measure was collected for only 150 in the Exparel arm and 135 in the Regular Bupivacaine group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exparel® | Regular Bupivacaine
Number analyzed (Participants) | 150 | 135
units on a scale | 4 (2.35) | 3.53 (3.6)
Statistical Analysis 1: Comparison: Exparel® vs Regular Bupivacaine; Test type: Superiority; p = 0.202, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Overall Opioid Use
Description: The total amount in mg of opioid medication consumed through 12, 24, 36, 48, 60, and 72 hours after surgery will be assessed.
Time Frame: Over the first 72 hours after surgery
Reporting Status: Not Posted

11. Secondary Outcome: Mean Length of Hospital Stay
Description: Indirect outcome measure to assess the adequacy of postoperative pain control as an indicator of improvement in healing period, patient participation in physical therapy and faster patient mobilization, and overall health care cost
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Change From Baseline in Quality of Life
Description: The impact of pain on patient's quality of life will be assessed through a brief pain inventory (BPI). In addition, the 5-point scale analgesia satisfaction survey will be used along with the BPI to assess patient satisfaction and quality of life.
Time Frame: Will be assessed preoperatively, on the first post-op day (POD 1), on POD2, and POD 3
Reporting Status: Not Posted

13. Secondary Outcome: Number of Participants Who Attain Physical Therapy Goal That Justifies Discharge From Inpatient Physical Therapy Within 72 Hours
Time Frame: 72 hours after surgery
Reporting Status: Not Posted

14. Secondary Outcome: Hospital Cost for Patient Care During Hospitalization
Description: Hospital cost for patient care during hospitalization will be estimated from hospital charges and financial records.
Time Frame: duration of hospital stay, an expected average of 4 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 days after surgery
Description: Only adverse events that were related to the study drug were collected.
Arm/Group | Exparel® | Regular Bupivacaine
All-Cause Mortality (participants affected / at risk) | 4/171 | 2/175
Serious Adverse Events (participants affected / at risk) | 0/171 | 0/175
Other Adverse Events (participants affected / at risk) | 0/171 | 0/175

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT02111746/Prot_SAP_002.pdf